CLINICAL TRIAL: NCT06348264
Title: Adjuvant Rezvilutamide in Combination With Androgen Deprivation Therapy in Androgen Receptor-positive, High-risk Salivary Duct Carcinoma: a Single-arm Phase 2 Trial
Brief Title: Adjuvant Rezvilutamide in Combination With Androgen Deprivation Therapy in Androgen Receptor-positive, High-risk Salivary Duct Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry); Beijing Biote Pharmaceutical Co.,Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDC-1
Record Dates: First submitted 2024-03-30; First posted 2024-04-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Salivary Gland Neoplasm Duct
MeSH Terms: interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rezvilutamide plus LHRHa (Experimental): Participants will receive rezvilutamide in combination with a LHRHa for up to 2 years.
  Interventions: Drug: Rezvilutamide; Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Rezvilutamide — Rezvilutamide 240 mg (3*80mg tablets) will be administered orally once daily with or without food.
Drug: Leuprolide Acetate — The dose and frequency of administration will be consistent with the prescribing information in prostate cancer patients.

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of rezvilutamide in combination with androgen deprivation therapy (ADT) in participants with androgen receptor (AR) positive, high-risk salivary duct carcinoma (SDC).

The procedures include screening, treatment and follow-up period. The treatment includes rezvilutamide plus Luteinizing Hormone Releasing Hormone agonist (LHRHa) for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Histologically confirmed salivary duct carcinoma and stage III or IVa or IVb according to AJCC Cancer Staging Manual Eighth Edition
* Completed SDC surgery, and adjuvant radiotherapy is planned or ongoing or has completed
* Androgen receptor (AR) positive
* White blood cell (WBC) ≥ 3.0 x 10^9/L, Neutrophil count≥ 1.5 x 10^9/L, Platelet count (PLT) ≥ 75 x 10^9/L, Haemoglobin (Hb) ≥ 90 g/L
* Serum creatinine (Cr) < 1.5 x upper limit of normal(ULN) or creatinine clearance ≥ 50 ml/min.
* Total bilirubin (TBIL) < 1.5 x ULN, AST< 2.5 x ULN, and ALT< 2.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2, and ability to take oral medication
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 1 year after the end of study intervention administration
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

* Received prior anti-AR pathway therapy
* Treatment with another investigational drug or chemotherapy within 6 months
* History of hypothalamus or pituitary dysfunction
* History of seizure
* Clinically uncontrolled diseases, such as septic shock, uncontrolled hypertension, unstable angina, New York Heart Association (NYHA) class III or IV heart disease, clinically unstable arrhythmia, myocardial infarction (in the past 6 months)
* Previous cancer except skin cancer rather than malignant melanoma or any cancer curatively treated > 5 years prior to study entry
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2031-03-30 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival (DFS) | 36 months
  DFS is defined as the time from entry until disease recurrence or death

SECONDARY OUTCOMES:
3-year overall survival (OS) | 36 months, 60 months
  OS is defined as the time from entry until death due to any cause
3-year disease-specific survival (DSS) | 36 months, 60 months
  DSS is defined as the time from entry until disease-specific death
3-year distant-metastatic free survival (DMFS) | 36 months, 60 months
  DMFS is defined as the time from entry until distant metastasis or death
Adverse events | 36 months
  Evaluate adverse events utilizing CTCAE V5
5-year disease-free survival (DFS) | 60 months
  DFS is defined as the time from entry until disease recurrence or death

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University School and Hospital of Stomatology, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No